CLINICAL TRIAL: NCT06979063
Title: Impact of Regulation Strategies and Health Education for Managing Infertility in Primary Health Care in Rio Grande do Sul
Brief Title: Health Education for Women With Suspeced Infertility Waiting for Specialized Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Telessaúde RS (Unknown)
Responsible Party: Principal Investigator, Michele Zschornack Strelow, Principal Investigator, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022-0588
Record Dates: First submitted 2025-04-24; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Infertility; Health Education; Telemedicine; Telehealth
MeSH Terms: conditions — Infertility; Health Education | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: This is an open-label, superiority, randomized controlled trial with two parallel groups. Participants will be assigned to either a control group, which follows standard care, or an intervention group, which receives remote counseling and education about infertility and healthcare system navigation.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor and the statistician will be masked to group allocation. All other participants, investigators, and care providers will be aware of the assigned intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): Wait for specialized infertility consultation, following the usual health system process.
  Interventions: Other: Standard Care Arm
- intervention group (Experimental): Remote counseling and education about infertility and healthcare system navigation.
  Interventions: Other: Remote Infertility Education and Counseling; Other: Standard Care Arm

INTERVENTIONS:
Other: Remote Infertility Education and Counseling — Patients receive video call counseling covering infertility investigation, non-pharmacological fertility enhancement strategies, and healthcare navigation guidance.
  Health professionals review patient records and request missing infertility-related exams according to local protocol.
  Additional follow-ups occur approximately every 30 days to assist with pending investigations.
  If significant findings arise, patients will receive an explanation and assistance in scheduling primary care consultations.
  Arms: intervention group
Other: Standard Care Arm — Referrals from patients will be avaluated following local protocols in the electronic referral system. Incomplete data will be requested through this system. There will be no direct contact with patients.

SUMMARY:
Introduction: Infertility is defined as a couple's inability to achieve pregnancy after 12 months or more of regular unprotected intercourse. In Brazil, it affects around eight million people. While health services provide resources for contraception, little attention is given to supporting conception and preserving fertility.

Objective: To evaluate the effectiveness of a remote educational and counseling intervention on infertility.

Method: Open-label randomized clinical trial. Couples referred for infertility will be identified in the electronic referral system. For inclusion, the woman of the couple must be 34 years old or less, no previous in-vitro fertilization attempts, and have access to telephone or internet. The control group will follow standard care, awaiting in-person consultation. The intervention group will also wait for in-person evaluation but receive additional education and counseling via video call.

The primary outcome is the proportion of correct referrals according to local protocols. A total of 206 participants will be included to detect a difference between success rates of 50% and 30%, with 80% power and a 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* Individuals referred to specialized infertility care in Porto Alegre.
* Age up to 33 years and 11 months.

Exclusion Criteria:

* Lack of access to the internet or telephone.
* Prior specialized infertility treatment in the private healthcare system.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Correct referral | Six months after randomization
  Proportion of participants correctly referred to specialized care according to local protocols.

SECONDARY OUTCOMES:
Proportion of patients with conception plan achieved. | Six months after randomization
  Patient-reported conception plan will be evaluated by interview to assess whether pregnancy was achieved or it was opted to forgo the plan.
FertiQoL | Six months after randomization
  Change in Quality of Life as Measured by the Fertility Quality of Life (FertiQoL) Questionnaire. The FertiQoL is a validated instrument that measures quality of life in individuals experiencing fertility problems. Scores range from 0 to 100, where higher scores indicate better quality of life.
Time to regulation decision | Six months after randomization
  Time in days between the referral and final decision for the referral
Time for in-person consulting | Six months after randomization
  Time in days between the referral and in-person consult.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided